CLINICAL TRIAL: NCT05951894
Title: Flow-mediated Arterial Dilatation, Hypertension, Endothelin-1 (ET-1) and Soluble Intercellular Adhesion Molecule (sICAM-1) in Obese Adolescents
Brief Title: Flow-mediated Arterial Dilatation, Hypertension, Endothelin-1 and sICAM-1 in Obese Adolescents
Acronym: sICAM-1
Status: Completed | Type: Observational
Sponsor: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Nur Aisiyah Widjaja, Principal Investigator on Nutrition and Metabolic Disease, Universitas Airlangga
Other Study IDs: A Number; UA number (Other: Airlangga University)
Record Dates: First submitted 2023-06-19; First posted 2023-07-19 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Hypertension; Adolescent Obesity
Keywords: Obesity; Flow-mediated Arterial Dilatation; Hypertension; sICAM-1
MeSH Terms: conditions — Obesity; Hypertension; Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Biospecimen Retention: Samples Without DNA — the samples in the form of blood for investigation: lipid profile, fasting blood glucose, fasting insulin, endothelin-1 adn sICAM-1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypertension: This group consists of obese adolescents with hypertension, defined as systole blood pressure >130 mmHg or diastole blood pressure >85 mmHg, or both
- Non-hypertension: This group consists of obese adolescents without hypertension
- Normal (non-obese): This group consist of normal subjects (non-obese)

SUMMARY:
Obesity in adolescents is associated with the development of cardiovascular disease and type 2 diabetes mellitus. In order to detect early development of cardiovascular disease, early detection of the endothelium of obese adolescents is needed. Endothelium dysfunction is an early stage of developing atherosclerosis, which can be a predictor of cardiovascular disease development in the future. Flow mediated dilatation (FMD) is a non-invasive method that can measure endothelium function and predict the risk of cardiovascular disease, which is not only able to measure artery diameter, but also provides function index of nitric oxide (NO) in the endothelium. FMD is negatively related to BMI. Meanwhile, Endothelin-1 (ET-1) is thought to play a role in the pathogenesis of insulin resistance, because when its levels increase, ET-1 can cause a condition of hyperinsulinemia. ET-1 was found to be high in patients with cardiovascular disorders, as well as in obese and diabetic subjects. Alternative methods for assessing endothelial function by measurement of biomarkers of activation and endothelial dysfunction such as soluble intercellular adhesion molecule-1 (sICAM-1). Levels of sICAM-1 have been found to be related positively to age, systolic and diastolic blood pressure, hypercholesterolemia, hypertriglyceridemia and inversely to estrogen. Furthermore, associations have been found between sICAM-1 and cardiovascular mortality in both healthy individuals and populations at high risk.

The aim of the study was to evaluate FMD, concentrations of ET-1 and sICAM-1 in adolescents with a presence of obesity and hypertension and to compare these with controls (obesity and non hypertension), as well as to analyze the correlations between FMD, ET-1, sICAM-1 and blood pressure values.

DETAILED DESCRIPTION:
This study is cross sectional study with observational analytic that evaluates FMD, ET-1 dan sICAM-1 in obese adolescents with hypertension compared to obese adolescents without hypertension and normal adolescents. The subjects are 70 adolescents (obese and normal) aged 13-18 years, healthy, not undergoing any medication, not smoking and not drinking alcohol, which are further divided into 3 groups: obesity with hypertension, obesity without hypertension and normal. Examination includes blood pressure examination, brachial ultrasound and blood sampling to measure levels of profile lipid, blood glucose, ET-1, and sICAM-1. Blood sample of subjects were taken by laboratory employee of the general hospital in Surabaja, Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Obesity
* Healthy
* Study in Junior or Senior High School in Surabaja city

Exclusion Criteria:

* Smoking or consuming alcohol
* Suffering from infections, inflammation, autoimmune diseases, cancer, chronic diseases, and endocrine disorders
* consuming steroids or hormone therapy

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Obese adolescents aged 13-18 years old
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Body height | 5 months
  Body height will be measured using Seca 213 stadiometer. The subjects were asked to step at the stadiometer base in an upright state, with the heel, the buttock, and the shoulder blade touching the scale pool. The chin up, look straight ahead. The head slider was lowered until it touches the cranium. Noted the body height in the data collection sheet (presenting in mean +/- SD, in cm). The subject must use light clothes without accessories or footwear, such as hats or hair ponytail.
Body weight | 5 months
  Body weight will be measured using Tanita RD 953-BK digital scale (presenting in mean +/- SD, in kg). The subjects were asked to step at the scale in an upright state. The body weight appears on the screen and is then noted in the data collection sheet. The subject must use light clothes without accessories or footwear
Hip circumference (HC) | 5 months
  Hip circumference will be measured using Seca 201 measuring tape (in cm), by asking the subjects to keep the feet together, then wrapping the measuring tape around the widest part of the hips, at the point of the greatest gluteal protuberance. The subjects were measured using light cloth without food wear and other accessories such as belts, hats, hair accessories, etc. The data will be presented as mean +/- SD
Waist circumference (WC) | 5 months
  Waist circumference will be measured using Seca 201 measuring tape (in cm), Waist circumference was measured by wrapping the measuring tape around the subject's stomach, at the midpoint between the lowest rib and the endpoint of the iliac crest upon expiration, in line with the navel. The subjects were measured using light cloth without food wear and other accessories such as belts, hats, hair accessories, etc. The data will be presented as mean +/- standard deviation (SD)
Flow-mediated Arterial Dilatation diameter | 5 months
  FMD was calculated as the maximum percentage increase in diameter of the brachial artery after ischemia of the forearm. The measurements were performed in supine position at the elbow of the right arm. The cuff was placed on the forearm, distally to the measurement site. The duration of ischemia of the forearm was 5 min. All lumen diameter measurements were done at end diastole by the use of the R-wave of the electrocardiogram. The ultrasound images were made by one technician with a 7.5 megahertz (MHz) linear array transducer of an Ultramark duplex scanner. All images were stored on flash-disk for off-line analysis. Measurement of the endothelium-independent vasodilatation using nitroglycerine, was not performed.
Endothelin-1 | 5 months
  Endothelin-1 will be analyzed using the Human Endothelin-1 Elisa kit (Bioassay Technology Laboratory) (in ng/ml). The data will be presented as mean +/- standard deviation (SD)
sICAM-1 | 5 months
  sICAM-1 will be analyzed using Human intercellular adhesion molecule 1 Elisa kit (Bioassay Technology Laboratory) (in ng/ml). The data will be presented as mean +/- standard deviation (SD)

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 5 months
  BMI was calculated by dividing body weight (in kg) by body height square (in m) [body weight (kg)/body height2 (m2)], in kg/m2 unit. The data will be presented as mean +/- standard deviation (SD)
Systolic blood pressure | 5 months
  Systolic blood pressure was measure using Omron Automatic Blood Pressure Monitor (Omron Health Care Co., Ltd, Japan) (in mmHg), by placing the cuff on the right arm, then pull and tighten it according to the size if the arm. After it was installed correctly (fasten and did not move), the power button on the digital tension tool was pressed, and then the microprocessor started to drive air pressure into the cuff, and then the value of blood pressures will appear in the manometer tube column. Systolic blood pressure measurement was performed in a sitting position after the subject had rested for 10 minutes. The data will be presented as mean +/- standard deviation (SD)
Diastolic blood pressure | 5 months
  Diastolic blood pressure was measure using Omron Automatic Blood Pressure Monitor (Omron Health Care Co., Ltd, Japan) (in mmHg), by placing the cuff on the right arm, then pull and tighten it according to the size if the arm. After it was installed correctly (fasten and did not move), the power button on the digital tension tool was pressed, and then the microprocessor started to drive air pressure into the cuff, and then the value of blood pressures will appear in the manometer tube column. Diastolic blood pressure measurement was performed in a sitting position after the subject had rested for 10 minutes. The data will be presented as mean +/- standard deviation (SD)
Fasting blood glucose | 5 months
  Blood samples were collected at 08.00-09.00 after the subject fasted for 12 hours through the median cubital vein. Ten ml of blood was taken. The blood sample collection was done by a laboratory's employers or a nurse who had been hired by the researchers. After the blood was taken, it was placed into a tube containing ethylenediaminetetraacetic acid (EDTA) for further analysis of fasting blood glucose (FBG). After that, the tube containing blood samples was placed in a cooling box for transport to the lab. The data will be presented as mean +/- SD, in mg/dL.
Total cholesterol | 5 months
  Blood samples were collected at 08.00-09.00 after the subject fasted for 12 hours through the median cubital vein. Ten ml of blood was taken. The blood sample collection was done by a laboratory's employers or a nurse who had been hired by the researchers. After the blood was taken, it was placed into a tube containing ethylenediaminetetraacetic acid (EDTA) for further analysis of Total cholesterol. After that, the tube containing blood samples was placed in a cooling box for transport to the lab. The data will be presented as mean +/- SD, in mg/dL.
HDL-c | 5 months
  Blood samples were collected at 08.00-09.00 after the subject fasted for 12 hours through the median cubital vein. Ten ml of blood was taken. The blood sample collection was done by a laboratory's employers or a nurse who had been hired by the researchers. After the blood was taken, it was placed into a tube containing ethylenediaminetetraacetic acid (EDTA) for further analysis of High-density lipoprotein cholesterol (HDL-c). After that, the tube containing blood samples was placed in a cooling box for transport to the lab. The data will be presented as mean +/- SD, in mg/dL.
LDL-c | 5 months
  Blood samples were collected at 08.00-09.00 after the subject fasted for 12 hours through the median cubital vein. Ten ml of blood was taken. The blood sample collection was done by a laboratory's employers or a nurse who had been hired by the researchers. After the blood was taken, it was placed into a tube containing ethylenediaminetetraacetic acid (EDTA) for further analysis of Low-density lipoprotein cholesterol (LDL-c). After that, the tube containing blood samples was placed in a cooling box for transport to the lab. The data will be presented as mean +/- SD, in mg/dL.
Triglyceride | 5 months
  Blood samples were collected at 08.00-09.00 after the subject fasted for 12 hours through the median cubital vein. Ten ml of blood was taken. The blood sample collection was done by a laboratory's employers or a nurse who had been hired by the researchers. After the blood was taken, it was placed into a tube containing ethylenediaminetetraacetic acid (EDTA) for further analysis of Triglycerides After that, the tube containing blood samples was placed in a cooling box for transport to the lab. The data will be presented as mean +/- SD, in mg/dL.
Fasting insulin | 5 months
  Blood samples were collected at 08.00-09.00 after the subject fasted for 12 hours through the median cubital vein. Ten ml of blood was taken. The blood sample collection was done by a laboratory's employers or a nurse who had been hired by the researchers. After the blood was taken, it was placed into a tube containing ethylenediaminetetraacetic acid (EDTA) for further analysis of Fasting insulin (FI). After that, the tube containing blood samples was placed in a cooling box for transport to the lab. The data will be presented as mean +/- SD, in μU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Budi Santoso, Professor, Study Chair — Universitas Airlangga; Achmad Tri Ludfy Avianto, MD, Study Chair — Universitas Airlangga
Locations (1):
- RS Bhayangkara Surabaya, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao W, Mo L, Pang Y. Hypertension in adolescents: The role of obesity and family history. J Clin Hypertens (Greenwich). 2021 Dec;23(12):2065-2070. doi: 10.1111/jch.14381. Epub 2021 Nov 16. PMID 34783422
- [Result] Koenen M, Hill MA, Cohen P, Sowers JR. Obesity, Adipose Tissue and Vascular Dysfunction. Circ Res. 2021 Apr 2;128(7):951-968. doi: 10.1161/CIRCRESAHA.121.318093. Epub 2021 Apr 1. PMID 33793327
- [Result] Bellamkonda K, Williams M, Handa A, Lee R. Flow Mediated Dilatation as a Biomarker in Vascular Surgery Research. J Atheroscler Thromb. 2017 Aug 1;24(8):779-787. doi: 10.5551/jat.40964. Epub 2017 Jul 1. PMID 28674324
- [Result] Weissgerber TL. Flow-mediated dilation: can new approaches provide greater mechanistic insight into vascular dysfunction in preeclampsia and other diseases? Curr Hypertens Rep. 2014 Nov;16(11):487. doi: 10.1007/s11906-014-0487-z. PMID 25182159
- [Result] Green DJ, Jones H, Thijssen D, Cable NT, Atkinson G. Flow-mediated dilation and cardiovascular event prediction: does nitric oxide matter? Hypertension. 2011 Mar;57(3):363-9. doi: 10.1161/HYPERTENSIONAHA.110.167015. Epub 2011 Jan 24. PMID 21263128
- [Result] Maruhashi T, Kajikawa M, Kishimoto S, Hashimoto H, Takaeko Y, Yamaji T, Harada T, Han Y, Aibara Y, Mohamad Yusoff F, Hidaka T, Kihara Y, Chayama K, Nakashima A, Goto C, Tomiyama H, Takase B, Kohro T, Suzuki T, Ishizu T, Ueda S, Yamazaki T, Furumoto T, Kario K, Inoue T, Koba S, Watanabe K, Takemoto Y, Hano T, Sata M, Ishibashi Y, Node K, Maemura K, Ohya Y, Furukawa T, Ito H, Ikeda H, Yamashina A, Higashi Y. Diagnostic Criteria of Flow-Mediated Vasodilation for Normal Endothelial Function and Nitroglycerin-Induced Vasodilation for Normal Vascular Smooth Muscle Function of the Brachial Artery. J Am Heart Assoc. 2020 Jan 21;9(2):e013915. doi: 10.1161/JAHA.119.013915. Epub 2020 Jan 8. PMID 31910779
- [Result] Jenkins HN, Rivera-Gonzalez O, Gibert Y, Speed JS. Endothelin-1 in the pathophysiology of obesity and insulin resistance. Obes Rev. 2020 Dec;21(12):e13086. doi: 10.1111/obr.13086. Epub 2020 Jul 6. PMID 32627269
- [Result] Yang L, Magnussen CG, Yang L, Bovet P, Xi B. Elevated Blood Pressure in Childhood or Adolescence and Cardiovascular Outcomes in Adulthood: A Systematic Review. Hypertension. 2020 Apr;75(4):948-955. doi: 10.1161/HYPERTENSIONAHA.119.14168. Epub 2020 Mar 2. PMID 32114851
- [Result] Dulskiene V, Kuciene R, Medzioniene J, Benetis R. Association between obesity and high blood pressure among Lithuanian adolescents: a cross-sectional study. Ital J Pediatr. 2014 Dec 10;40:102. doi: 10.1186/s13052-014-0102-6. PMID 25492217
- [Result] Widjaja NA, Irawan R, Prihaningtyas RA, Ardiana M, Hanindita MH. Carotid intima-media thickness, hypertension, and dyslipidemia in obese adolescents. Pan Afr Med J. 2019 Nov 7;34:134. doi: 10.11604/pamj.2019.34.134.18309. eCollection 2019. PMID 33708303
- [Result] Rundek T, Gardener H, Della-Morte D, Dong C, Cabral D, Tiozzo E, Roberts E, Crisby M, Cheung K, Demmer R, Elkind MS, Sacco RL, Desvarieux M. The relationship between carotid intima-media thickness and carotid plaque in the Northern Manhattan Study. Atherosclerosis. 2015 Aug;241(2):364-70. doi: 10.1016/j.atherosclerosis.2015.05.027. Epub 2015 Jun 3. PMID 26071659
- [Result] Rivera-Gonzalez O, Wilson NA, Coats LE, Taylor EB, Speed JS. Endothelin receptor antagonism improves glucose handling, dyslipidemia, and adipose tissue inflammation in obese mice. Clin Sci (Lond). 2021 Jul 30;135(14):1773-1789. doi: 10.1042/CS20210549. PMID 34278410
- [Result] Busjahn A, Knoblauch H, Knoblauch M, Bohlender J, Menz M, Faulhaber HD, Becker A, Schuster H, Luft FC. Angiotensin-converting enzyme and angiotensinogen gene polymorphisms, plasma levels, cardiac dimensions. A twin study. Hypertension. 1997 Jan;29(1 Pt 2):165-70. doi: 10.1161/01.hyp.29.1.165. PMID 9039097
- [Result] Giannini C, de Giorgis T, Scarinci A, Cataldo I, Marcovecchio ML, Chiarelli F, Mohn A. Increased carotid intima-media thickness in pre-pubertal children with constitutional leanness and severe obesity: the speculative role of insulin sensitivity, oxidant status, and chronic inflammation. Eur J Endocrinol. 2009 Jul;161(1):73-80. doi: 10.1530/EJE-09-0042. Epub 2009 May 7. PMID 19423560
- [Result] Witte DR, Broekmans WM, Kardinaal AF, Klopping-Ketelaars IA, van Poppel G, Bots ML, Kluft C, Princen JM. Soluble intercellular adhesion molecule 1 and flow-mediated dilatation are related to the estimated risk of coronary heart disease independently from each other. Atherosclerosis. 2003 Sep;170(1):147-53. doi: 10.1016/s0021-9150(03)00253-3. PMID 12957693
- [Result] Dzikowska-Diduch O, Domienik-Karlowicz J, Gorska E, Demkow U, Pruszczyk P, Kostrubiec M. E-selectin and sICAM-1, biomarkers of endothelial function, predict recurrence of venous thromboembolism. Thromb Res. 2017 Sep;157:173-180. doi: 10.1016/j.thromres.2017.07.027. Epub 2017 Jul 26. PMID 28780342
- [Result] Glowinska B, Urban M, Peczynska J, Florys B. Soluble adhesion molecules (sICAM-1, sVCAM-1) and selectins (sE selectin, sP selectin, sL selectin) levels in children and adolescents with obesity, hypertension, and diabetes. Metabolism. 2005 Aug;54(8):1020-6. doi: 10.1016/j.metabol.2005.03.004. PMID 16092051